CLINICAL TRIAL: NCT05532124
Title: LAENNEC (Human Placenta Hydrolysate) Stiffness of Chronic Liver Disease Patients to Evaluate the Safety and Effectiveness of Multi -Tube, Eye, Placebo, and Capacity Increase and Capacity Enlargement Clinical Trial to Assess the Safety and Effectiveness
Brief Title: Part A: In Patients With Chronic Liver Diseases, LAENNEC (Human Placenta Hydrolysate) is to Assess Safety and Tolerability After the Doses of Doses. Part B: Part A, it is to Determine the Optimal Dose by Evaluating Two Capacity and Placebo Groups.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Wellbeing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAEN-IV2A
Record Dates: First submitted 2022-09-01; First posted 2022-09-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-09

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A: LAENNEC 4ml (Experimental): Dosing twice a week for 2 weeks
  Interventions: Biological: LAENNEC (Human Placenta Hydrolysate)
- Part A: LAENNEC 6ml (Experimental): Dosing twice a week for 2 weeks
  Interventions: Biological: LAENNEC (Human Placenta Hydrolysate)
- Part A: LAENNEC 10ml (Experimental): Dosing twice a week for 2 weeks
  Interventions: Biological: LAENNEC (Human Placenta Hydrolysate)
- Part A: Normal Saline (Active Comparator): Dosing twice a week for 2 weeks
  Interventions: Other: normal saline
- Part B: LAENNEC 1 (Experimental): It is administered twice a week or placebo, and administered until it is normalized for up to 6 weeks or ALT.
  Interventions: Biological: LAENNEC (Human Placenta Hydrolysate)
- Part B: LAENNEC 2 (Experimental): It is administered twice a week or placebo, and administered until it is normalized for up to 6 weeks or ALT.
  Interventions: Biological: LAENNEC (Human Placenta Hydrolysate)
- Part B: Normal Saline (Active Comparator): It is administered twice a week or placebo, and administered until it is normalized for up to 6 weeks or ALT.
  Interventions: Other: normal saline

INTERVENTIONS:
Biological: LAENNEC (Human Placenta Hydrolysate) — Intravenous Injection
  Arms: Part A: LAENNEC 10ml; Part A: LAENNEC 4ml; Part A: LAENNEC 6ml; Part B: LAENNEC 1; Part B: LAENNEC 2
Other: normal saline — Intravenous Injection
  Arms: Part A: Normal Saline; Part B: Normal Saline

SUMMARY:
Part A: In Patients With Chronic Liver Diseases, LAENNEC (Human Placenta Hydrolysate) is to Assess Safety and Tolerability After the Doses of Doses.

Part B: Part A, it is to Determine the Optimal Dose by Evaluating Two Capacity and Placebo Groups.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of screening, 18 or 75 years
2. Those who have been diagnosed with alcoholic or non -alcoholic fatty liver disease and have persisted for more than 6 months
3. Those who are 1.5 times (60 IU/L) of the ALT level of Baseline (60 IU/L)
4. A person who can complete the signature agreement and compliance the requirements for clinical trials.

Exclusion Criteria:

1. Liver function abnormalities caused by the following cause disease: viral hepatitis, biliary obstructions, autoimmune hepatitis, wilson disease, hematoprive
2. Drug allergic symptoms (oscillation, heat, itching)
3. Those with systemic infection (including tuberculosis)
4. If the test person judges that it is difficult to participate in clinical trials due to the next disease: Cirrhosis of CHILD C or higher, cirrhosis with edema and plural, malignant tumors, severe disorders, severe renal disorders, severe cardiovascular disease, severe nerve Mental disorders, preferences, etc.
5. Those who have experienced use of human -derived medicines within 6 months before selecting a test subject
6. Those who have received other clinical drugs within 3 months before selecting a test subject
7. Magnetic Resonance Spectroscopy (MRS) is impossible
8. A person who does not perform appropriate contraception as a pregnant woman, a nursing or a woman of childbearing age (effective contraception method: Barrier methods using infertility surgery, uterine device, condom, killer)
9. Those who cannot inject intravenous infusions
10. Those who judged that other testors were inappropriate as clinical trials

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
PartA: Adverse Event and clinical trials test | week 2
  The ratio of the test subjects who have experienced more than one Adverse Event is compared with the Chi-Square Test or Fisher's Exact Test.
  For clinical trial tests, the amount of change in the group is paired T-test, and the amount of changes between the groups is conducted with Independent Two Sample T-Test.
  Mcnemar 's Test is performed for normal and abnormal changes in the administration of clinical trial tests, and the difference between the divisions between the group is performed with the Generalized Estimating Equation (GEE).
PartB: Change amoust of ALT | week 6
  The ALT improvement rate of the test group and the control group is presented. The ALT proposes a ratio of test subjects that decreased by more than 20% compared to the base value, and compares the difference between the group using the Chi-Square Test or Fisher's Exact Test.

SECONDARY OUTCOMES:
PartA: Change amoust of ALT | week 2, 4 and 6
  The ALT improvement rate of the test group and the control group is presented. The ALT proposes a ratio of test subjects that decreased by more than 20% compared to the base value, and compares the difference between the group using the Chi-Square Test or Fisher's Exact Test.
PartA: Adverse Event and clinical trials test | week 6
  The ratio of the test subjects who have experienced more than one Adverse Event is compared with the Chi-Square Test or Fisher's Exact Test.
  For clinical trial tests, the amount of change in the group is paired T-test, and the amount of changes between the groups is conducted with Independent Two Sample T-Test.
  Mcnemar 's Test is performed for normal and abnormal changes in the administration of clinical trial tests, and the difference between the divisions between the group is performed with the Generalized Estimating Equation (GEE).
PartB: Adverse Event and clinical trials test | week 6
  The ratio of the test subjects who have experienced more than one Adverse Event is compared with the Chi-Square Test or Fisher's Exact Test.
  For clinical trial tests, the amount of change in the group is paired T-test, and the amount of changes between the groups is conducted with Independent Two Sample T-Test.
  Mcnemar 's Test is performed for normal and abnormal changes in the administration of clinical trial tests, and the difference between the divisions between the group is performed with the Generalized Estimating Equation (GEE).
PartB: Major liver function test (ALT, AST, γ-GT, total bilirubin) | week 2, 4 and 6
  Change amoust of ALT, AST, γ-GT, total bilirubin.
  Independent Two Sample T-Test compares the difference between the group

OTHER OUTCOMES:
PartA: Fat liver decrease effect (MRS) | week 6
  Absolute change from baseline in mean liver fat (MRS)
  Independent Two Sample T-Test compares the difference between the group
PartB: Fat liver decrease effect (MRS) | week 6
  Absolute change from baseline in mean liver fat (MRS)
  Independent Two Sample T-Test compares the difference between the group

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Keimyung university dongsan medical center, Daegu
  - Yeungnam university, Daegu
  - Hanyang University Hospital., Seoul
  - Korea university guro hospital, Seoul
  - Severance hospital, Seoul
  - Soonchunhyang university hospital, Seoul
  - Wonju severance christian hospital, Wŏnju